CLINICAL TRIAL: NCT04489524
Title: A Feasibility Study of Culturally Tailored Smoking Cessation for Chinese Smokers in New York City
Brief Title: Smoking Cessation in NYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Quit Smoking; U01CA114582-02S2 (NIH)
Record Dates: First submitted 2020-07-16; First posted 2020-07-28 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individualized counselor-led MI sessions and NRT (Experimental): The intervention (4 individualized counselor-led MI sessions and nicotine replacement therapy [NRT]) consisted of four 60-min in-person sessions of AMI counseling and a packet of self-help smoking cessation materials. Participants were provided NRT packs and counseled on their use.
  Interventions: Behavioral: individualized counselor-led MI sessions; Behavioral: NRT
- general health education, self-help materials, and NRT (Active Comparator): Participants in this condition were provided with four in-person 60-min health education sessions and packets of general health self-help information, nutrition, exercise, and the harmful effects of tobacco. Strategies for quitting smoking were also provided to participants in this group as well as a supply of NRT and counseling on its use.
  Interventions: Behavioral: general health education session; Behavioral: NRT

INTERVENTIONS:
Behavioral: individualized counselor-led MI sessions — Intervention consisted of four 60-min in-person sessions of AMI counseling and a packet of self help smoking cessation materials.
  Arms: individualized counselor-led MI sessions and NRT
Behavioral: general health education session — four in-person 60-min health education sessions and packets of general health self-help information, nutrition, exercise, and the harmful effects of tobacco.
  Arms: general health education, self-help materials, and NRT
Behavioral: NRT — nicotine replacement therapy

SUMMARY:
The investigators tested the feasibility of a culturally and linguistically sensitive smoking cessation program with combined counseling and pharmacological components for Chinese smokers in New York City; identified factors and techniques that enhance the administration and appropriateness of the intervention program; and examined the effectiveness of this program on quit attempts, quit rates, and overall smoking reduction.

ELIGIBILITY:
Inclusion Criteria:

* Primary eligibility criterion for inclusion in the study cohort was current smoking status. Other inclusion criteria were:

  1. self-identification as ethnic Chinese,
  2. aged 18 years and older,
  3. having smoked or puffed on a cigarette during the previous week,
  4. willingness to participate in the smoking cessation study,
  5. access to a functional telephone,
  6. expected presence in the study geographic area for a year or more, and
  7. not having been enrolled in the past or at the current time in any smoking cessation treatment programs.

Exclusion Criteria:

1. being currently pregnant and
2. having had a recent diagnosis of cardiovascular disease.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

PRIMARY OUTCOMES:
change in smoking behavior | baseline, 1 week, 1, 3, and 6-month
  participants were asked whether they had smoked or had a puff on a cigarette and the number of cigarettes smoked in the past 7 days at multiple assessment points.
change in Carbon monoxide (CO) concentration | baseline, 6-month follow-up
  CO, a biomarker of smoking status, was assessed at baseline and 6-m follow up
change in the stages of smoking cessation | baseline, 1 week, 1, 3, and 6-month
  According to Prochaska and DiClemente ' s Stages of Change model, the stages are: precontemplation, contemplation, preparation, action, and maintenance. It's an ordinal variable that measured at multiple assessment points

CONTACTS AND LOCATIONS:
Overall Officials: Grace X Ma, PhD, Principal Investigator — Temple University
Locations (1):
- Center for Asian Health, Lewis Katz School of Medicine, Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Wu D, Ma GX, Zhou K, Zhou D, Liu A, Poon AN. The effect of a culturally tailored smoking cessation for Chinese American smokers. Nicotine Tob Res. 2009 Dec;11(12):1448-57. doi: 10.1093/ntr/ntp159. Epub 2009 Nov 13. PMID 19915080